CLINICAL TRIAL: NCT02994823
Title: The "Pooling" Expressed Breast Milk: A Method for Improving the Nutritional Intake of Premature Infants
Acronym: POOL-BM
Status: Terminated | Type: Observational
Why Stopped: prolonged device failure after just 10 participants and too long to resume
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: POOL-BM
Record Dates: First submitted 2016-09-02; First posted 2016-12-16 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Breastfeeding Mothers of Infants Hospitalized

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators compared a pooled mother's expressed breastmilk for 24 hours with individual pump session collection of milk to provide a more consistent caloric product without increasing bacterial contamination.

ELIGIBILITY:
Inclusion Criteria:

* Mother of newborn hospitalized in intensive care unit
* Mother using a breast pump in the unit and / or at home
* Mother respected the rules of handling and transport breastmilk
* No opposition mother

Exclusion Criteria:

* refusal

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Breastfeeding mothers of infants hospitalized
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
caloric value of breastmilk | at the end of each 24 hours collection from inclusion to the end of collection during 4 days
  The caloric value will be compared between the two groups (pooled expressed breastmilk versus individual expressed breastmilk)

SECONDARY OUTCOMES:
bacterial contamination of breastmilk | at the end of each 24 hours collection from inclusion to the end of collection during 4 days
  The bacterial contamination of breastmilk will be compared between the two groups with the value for colony-forming units per milliliter (cfu/mL) after plating on sheep blood agar and Chapman's agar.

CONTACTS AND LOCATIONS:
Overall Officials: Murielle Dobrzynski, Study Director — CHRU de Brest
Locations (1):
- CHUR de Brest, Brest, France